CLINICAL TRIAL: NCT02587273
Title: The Pharmacokinetics of Fentanyl in Intensive Care Patients
Acronym: FENTANYL06
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University of California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FENTANYL06. Version 8; 2006-000885-35 (EudraCT Number)
Record Dates: First submitted 2015-06-03; First posted 2015-10-27 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Multiple Organ Failure; Critical Care; Intensive Care
Keywords: Critical care; Intensive Care; Fentanyl; Pharmacokinetics; Multiple Organ Failure
MeSH Terms: conditions — Multiple Organ Failure | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fentanyl (Other): This is a pharmacokinetics study with a single arm. All participants will will undergo the intervention described under the intervention section
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — In this study there will be no administration of an investigational product per study protocol. The dosage of fentanyl will be according to the ICU's established procedures and the treating physician's judgment. The specific dose of fentanyl given to each patient will differ extensively. By routine, the ICU's in our hospital usually dose the fentanyl infusion as 0,5 - 6 μg/kg/hrs (kg = Ideal Body Weight). The intervention in this study will be a per protocol cessation in administration of fentanyl over a 6 hours period. Arterial blood samples, urine samples, pre and post filter samples and samples from dialysate will be collected during this 6 hours. If the patient needs opioid analgesia during the period, alternative opioid analgesia will be given.
  Other Names: Fentanyl Citrate

SUMMARY:
This study is part of a project intended to develop guidelines to optimise the dosing of fentanyl in intensive care patients.

This study will focus on determining:

* Whether the pharmacokinetics of fentanyl change during the ICU stay.
* To what extent / the degree of change in fentanyl pharmacokinetics in ICU patients.
* Which factors (e.g. physiological variables) that cause such a change.
* Based on simulations, determine context-sensitive half-times of fentanyl in ICU patients.

DETAILED DESCRIPTION:
Background:

Patients admitted to the Intensive Care Unit (ICU) for treatment involving mechanical ventilation will be in need of sedation and analgesia in order to relieve pain and discomfort from necessary therapeutic procedures (1-7). The opioid fentanyl is frequently used as part of these sedation regimens(1-7).

The pharmacokinetics (PK) and pharmacodynamics (PD) of fentanyl after long-term administration in ICU patients has not been studied extensively. In a study in children (fentanyl infusion time 7-144 hrs.), increased volume of distribution was found when compared to data obtained after short-term use (9). The volume of distribution of alfentanil was increased when compared with data obtained after short-term use in a study of adult ICU patients sedated with propofol and alfentanil (a rapid-onset opioid) for 24 hrs. post-operatively (10). A similar increase in distribution volume of another opioid, sufentanil, was found in adult ICU patients (average sufentanil infusion time 12 days)(11).

Experience obtained during clinical anaesthesia suggests that the duration of action in fentanyl is significantly prolonged after long-term intravenous infusions (12-13). This property of fentanyl seems to be caused by a combination of factors. Since fentanyl has a large volume of distribution there will be a continuous return of the drug from peripheral tissues, and the concentration of fentanyl in plasma will be maintained in a clinically active range for some time after a fentanyl infusion has been terminated (9). Fentanyl also potentiates the sedative effects of e.g. propofol and midazolam which contributes to a further protraction of the wake-up time (14-15).

In ICU patients these undesirable effects of fentanyl will probably be amplified as a result of major changes in volume of distribution and administration of fentanyl infusions for extensive periods of time (weeks). The investigators believe that knowledge of the PK of fentanyl in this population will be valuable to help designing optimised infusion regimens of fentanyl in the clinical setting of the ICU.

Study Objective:

The main study objective is to determine wether the pharmacokinetics of fentanyl change during the ICU stay, and the extent of this change. The investigators will try to unveil which factors (e.g physiological variables) that cause such change, and based on simulations, determine context-sensitive half-times of fentanyl in ICU patients. As a result of this study the investigators aim to develop an infusion pump program to predict fentanyl plasma concentrations, and the recovery time of fentanyl effect (time to plasma concentration 1 ng/ml). Furthermore the investigators intend to test if the fentanyl infusion pump program predicts fentanyl plasma concentrations in a separate group of ICU patients.

Study Procedures:

In this study there will not be administration of an investigational product per study protocol. The dosage and administration of fentanyl will be according to the ICUs established procedures and the treating physician's judgment of what is appropriate for the patient. In the ICUs of Oslo University Hospital fentanyl is administered intravenously as a continuous infusion on an infusion pump System or if needed as single bolus doses given by a handheld syringe. By routine ICUs in Oslo University Hospital usually dose the fentanyl infusion as 0,5 - 6 μg/kg/hrs, where kg is a calculation of the patients Ideal Body Weight. The fentanyl used is from marketed stock in the ICUs and is delivered by the hospital pharmacy. All medication is labelled with information and stored according to local regulations. Participants will be recruited from surgical, neurosurgical and medical ICUs.

On study days the investigator will screen the patients admitted to the ICU during the last 24 hrs. If patients are eligible for the study due to the selection criteria, they will be included in a chronological order.

Each subject must give his/hers informed consent. The gravity of the clinical situation for ICU patients may preclude informed consent before inclusion in the study. In that case, the patient's relatives (or legal representative) will receive information about the study, and will be provided the opportunity to express their opinion. If the patient´s relatives (or legal representative) are against participation, the patient will not be included.

Daily sedation cessation and spontaneous awakening trials are implemented as standard treatment regimens in the ICU's of Oslo University Hospital. In this study the investigators intend to collect blood samples over a sedation cessation period, when no fentanyl is to be administered to the patient. If the participants needs opioid analgesia during this period, alternative opioid painkillers will be given.

The first blood sample will be collected right before administration of fentanyl is to be temporarily stopped. During the following hours repeated samples will be collected. The samples will be collected randomly within a time block containing consecutive time points. Each participant will accordingly contribute samples from the entire collection time period. Fentanyl will again be given as prescribed by the treating physician when the sedation cessation period has ended.

Samples will be spinned and stored on ice in a biobank for later analysis at The Dept. of Clinical Pharmacology, St.Olavs Hospital, Trondheim, Norway.

If participants in the study undergo treatment with continuous veno venous haemodialysis (CVVHD), investigators want to assess whether haemodialysis influences the degree of change in fentanyl PK. Haemodialysis is thought to have minimal effect upon the clearance of fentanyl, since fentanyl is mostly cleared by non-renal mechanisms. In addition fentanyl has high molecular weight, high protein binding capacity, low water solubility and an abundant volume of distribution that make it less likely dialyzable (16-17). There will be collected blood samples from the prefilter and postfilter line of the hemodialysis machine to asses if the dialysis filter might absorb fentanyl and remove drug from the circulation. The sampling times will follow the predefined block-sampling regimen of the arterial blood tests. Investigators also plan to calculate dialysis clearance of fentanyl in a subset of 10 patients.

Fentanyl is primarily metabolized in the liver by the Cytochrome P450 3A (CYP3A) enzymatic route (18-19). A study of genetic markers and polymorphism in the genes coding for these enzymes could possibly explain some of the variation in fentanyl PK in the ICU population (20-21). There will be collected a blood sample for later DNA processing to search for relevant genetic markers and polymorphisms in Cytochrome P450 enzymes.

The main metabolite of fentanyl is norfentanyl (18-19). Concentration of norfentanyl in the daily arterial blood samples will be quantified to make it possible to calculate the metabolic ratio of fentanyl/norfentanyl. The metabolic ratio will indicate to which extent each participant metabolizes fentanyl without having to take the plasma concentrations into account.

Norfentanyl is eliminated by the kidneys(18-19). There will be taken daily samples of urine to determine the urine concentrations of this metabolite.

To further asses possible covariates of fentanyl PK, patient demographics, medical history, co-morbidity, data descriptive of the population, concomitant medication and daily registrations of organ function parameters will be recorded for each patient during the study period.

Assessments and blood sampling will continue as long as the patient needs artificial ventilation and are treated with significant amounts of fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted to the ICU at Oslo University Hospital - Ullevål, in whom mechanical ventilation for > 72 hrs. is expected
* Aged 18 - 80 years, both inclusive
* Serum beta-HCG negative if female of childbearing potential, aged 18 - 45 years (both inclusive)

Exclusion Criteria:

* Tracheally intubated > 12 hrs. before admittance to the ICU
* Known hypersensitivity to fentanyl or other opioids
* Post partum < 6 weeks and/or lactating
* Informed consent not received
* Any reason why, in the opinion of the investigator and/or the treating physicians, the patient should not participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Concentration versus time of fentanyl in plasma | Daily samples during a time frame of 360 min. as long as the participant needs artificial ventilation and fentanyl.
  Randomly collected time points within a time block of 7 consecutive time points post stop in daily fentanyl administration. Time blocks: Block1:0, 2,15, 45,120, 240, 360 min. Block2: 0, 4, 20, 60, 150, 270, 360 min. Block3: 0, 8, 25, 75, 180, 300, 360 min. Block4: 0, 10, 30, 90, 210, 330, 360 min.

SECONDARY OUTCOMES:
Concentrations of fentanyl and norfentanyl in urine | 1 daily sample as long as the participant needs artificial ventilation and are treated with fentanyl.
  Daily Sample from urine collected over 0 - 360 min. post stop in fentanyl administration.
Concentration versus time of fentanyl in plasma from sample pre-dialysis filter line | Daily samples during a time frame of 360 min. as long as the participant receives CVVH, artificial ventilation and fentanyl.
  Samples are collected at the same timepoints as the samples from the arterial line described in outcome 1.
Concentration versus time of fentanyl in plasma from sample at post-dialysis filter line | Daily samples during a time frame of 360 min. as long as the participant receives CVVH, artificial ventilation and fentanyl.
  Samples are collected at the same timepoints as the samples from the arterial line described in outcome 1.
Concentration of fentanyl in dialysate | 1 daily sample from dialysate in 10 participants receiving CVVH, artificial ventilation and are treated with fentanyl.
  Sample from dialysate collected over 0 - 360 min. post stop in fentanyl administration.
Concentration versus time of norfentanyl in plasma | Daily samples during a time frame of 360 min. as long as the participant needs artificial ventilation and fentanyl.
  Samples are collected in time blocks from the arterial line described in outcome 1.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Heier, Professor, Principal Investigator — Dept. of Anaesthesia, Oslo University Hospital
Locations (1):
- Oslo University Hospital, Ullevål, Oslo, Oslo County, Norway

REFERENCES:
- [Background] Liu LL, Gropper MA. Postoperative analgesia and sedation in the adult intensive care unit: a guide to drug selection. Drugs. 2003;63(8):755-67. doi: 10.2165/00003495-200363080-00003. PMID 12662124
- [Background] Wagner BK, O'Hara DA. Pharmacokinetics and pharmacodynamics of sedatives and analgesics in the treatment of agitated critically ill patients. Clin Pharmacokinet. 1997 Dec;33(6):426-53. doi: 10.2165/00003088-199733060-00003. PMID 9435992
- [Background] Gehlbach BK, Kress JP. Sedation in the intensive care unit. Curr Opin Crit Care. 2002 Aug;8(4):290-8. doi: 10.1097/00075198-200208000-00004. PMID 12386488
- [Background] Hogarth DK, Hall J. Management of sedation in mechanically ventilated patients. Curr Opin Crit Care. 2004 Feb;10(1):40-6. doi: 10.1097/00075198-200402000-00007. PMID 15166848
- [Background] Patel SB, Kress JP. Sedation and analgesia in the mechanically ventilated patient. Am J Respir Crit Care Med. 2012 Mar 1;185(5):486-97. doi: 10.1164/rccm.201102-0273CI. Epub 2011 Oct 20. PMID 22016443
- [Background] Puntillo KA, Arai S, Cohen NH, Gropper MA, Neuhaus J, Paul SM, Miaskowski C. Symptoms experienced by intensive care unit patients at high risk of dying. Crit Care Med. 2010 Nov;38(11):2155-60. doi: 10.1097/CCM.0b013e3181f267ee. PMID 20711069
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Fukuda K. Intravenous opioid anesthetics. In Anesthesia, 6th Ed (ed Miller RD), Elsevier Churchill Livingstone, Philadelphia, pp 379-437
- [Background] Katz R, Kelly HW. Pharmacokinetics of continuous infusions of fentanyl in critically ill children. Crit Care Med. 1993 Jul;21(7):995-1000. doi: 10.1097/00003246-199307000-00012. PMID 8319480
- [Background] Frenkel C, Schuttler J, Ihmsen H, Heye H, Rommelsheim K. Pharmacokinetics and pharmacodynamics of propofol/alfentanil infusions for sedation in ICU patients. Intensive Care Med. 1995 Dec;21(12):981-8. doi: 10.1007/BF01700659. PMID 8750122
- [Background] Ethuin F, Boudaoud S, Leblanc I, Troje C, Marie O, Levron JC, Le Moing JP, Assoune P, Eurin B, Jacob L. Pharmacokinetics of long-term sufentanil infusion for sedation in ICU patients. Intensive Care Med. 2003 Nov;29(11):1916-20. doi: 10.1007/s00134-003-1920-y. Epub 2003 Aug 16. PMID 12923616
- [Background] Hughes MA, Glass PS, Jacobs JR. Context-sensitive half-time in multicompartment pharmacokinetic models for intravenous anesthetic drugs. Anesthesiology. 1992 Mar;76(3):334-41. doi: 10.1097/00000542-199203000-00003. PMID 1539843
- [Background] Shafer SL, Varvel JR. Pharmacokinetics, pharmacodynamics, and rational opioid selection. Anesthesiology. 1991 Jan;74(1):53-63. doi: 10.1097/00000542-199101000-00010. PMID 1824743
- [Background] Vuyk J, Mertens MJ, Olofsen E, Burm AG, Bovill JG. Propofol anesthesia and rational opioid selection: determination of optimal EC50-EC95 propofol-opioid concentrations that assure adequate anesthesia and a rapid return of consciousness. Anesthesiology. 1997 Dec;87(6):1549-62. doi: 10.1097/00000542-199712000-00033. No abstract available. PMID 9416739
- [Background] Ourahma S, Marchetti F, Clergue F, Levron JC, Le Moing JP, Viars P. [Peroperative perfusion of fentanyl or sufentanil: plasma concentrations and postoperative respiratory changes]. Ann Fr Anesth Reanim. 1993;12(4):357-64. doi: 10.1016/s0750-7658(05)80101-7. French. PMID 8273922
- [Background] Dean M. Opioids in renal failure and dialysis patients. J Pain Symptom Manage. 2004 Nov;28(5):497-504. doi: 10.1016/j.jpainsymman.2004.02.021. PMID 15504625
- [Background] Joh J, Sila MK, Bastani B. Nondialyzability of fentanyl with high-efficiency and high-flux membranes. Anesth Analg. 1998 Feb;86(2):447. doi: 10.1097/00000539-199802000-00049. No abstract available. PMID 9459269
- [Background] Feierman DE, Lasker JM. Metabolism of fentanyl, a synthetic opioid analgesic, by human liver microsomes. Role of CYP3A4. Drug Metab Dispos. 1996 Sep;24(9):932-9. PMID 8886601
- [Background] Labroo RB, Paine MF, Thummel KE, Kharasch ED. Fentanyl metabolism by human hepatic and intestinal cytochrome P450 3A4: implications for interindividual variability in disposition, efficacy, and drug interactions. Drug Metab Dispos. 1997 Sep;25(9):1072-80. PMID 9311623
- [Background] Kuehl P, Zhang J, Lin Y, Lamba J, Assem M, Schuetz J, Watkins PB, Daly A, Wrighton SA, Hall SD, Maurel P, Relling M, Brimer C, Yasuda K, Venkataramanan R, Strom S, Thummel K, Boguski MS, Schuetz E. Sequence diversity in CYP3A promoters and characterization of the genetic basis of polymorphic CYP3A5 expression. Nat Genet. 2001 Apr;27(4):383-91. doi: 10.1038/86882. PMID 11279519
- [Background] Takashina Y, Naito T, Mino Y, Yagi T, Ohnishi K, Kawakami J. Impact of CYP3A5 and ABCB1 gene polymorphisms on fentanyl pharmacokinetics and clinical responses in cancer patients undergoing conversion to a transdermal system. Drug Metab Pharmacokinet. 2012;27(4):414-21. doi: 10.2133/dmpk.dmpk-11-rg-134. Epub 2012 Jan 24. PMID 22277678
- [Background] Wright PM. Population based pharmacokinetic analysis: why do we need it; what is it; and what has it told us about anaesthetics? Br J Anaesth. 1998 Apr;80(4):488-501. doi: 10.1093/bja/80.4.488. No abstract available. PMID 9640156
- [Background] Segredo V, Caldwell JE, Wright PM, Sharma ML, Gruenke LD, Miller RD. Do the pharmacokinetics of vecuronium change during prolonged administration in critically ill patients? Br J Anaesth. 1998 Jun;80(6):715-9. doi: 10.1093/bja/80.6.715. PMID 9771295